CLINICAL TRIAL: NCT03554889
Title: A Phase I Trial of Combined Nimotuzumab With NK Cells Adoptive Transfer for the Treatment of Advanced Cancer
Brief Title: Immunotherapy of Advanced Cancer Using a Combination Nimotuzumab and NK Cells
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hangzhou Cancer Hospital (Other)
Collaborators: Shanghai bokang bioengineering co., LTD (Unknown)
Responsible Party: Principal Investigator, Shixiu Wu, President of Hangzhou Cancer Hospital, Hangzhou Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HangzhouCH11
Record Dates: First submitted 2018-05-24; First posted 2018-06-13 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Advanced Cancer; ADCC; NK Cell Mediated Immunity; Nimotuzumab; Adaptive Transfer
MeSH Terms: interventions — nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Peripheral blood lymphocytes will be collected. The NK cell will be selected and expanded ex vivo, then adaptive transfer back into patients. A total of 5.0 x 10^8/L NK cells will be infused in one cycle.To avoid allergic reactions, 50 mg hydrocortisone was intramuscularly injected into patient 30 min before cells infusion every time. Best supportive care was also provided for patients. Nimotuzumab will be used 24 hours before infusion. Patients continued receiving treatment unless they had unacceptable adverse effects, or progressive disease confirmed by CT and PET-CT or they withdrew consent.
  Interventions: Biological: NK Cell adaptive transfer; Drug: Nimotuzumab

INTERVENTIONS:
Biological: NK Cell adaptive transfer — Nimotuzumab will enhance the ADCC effect of NK Cell adaptive transfer
Drug: Nimotuzumab — Nimotuzumab will enhance the ADCC effect of NK Cell adaptive transfer

SUMMARY:
NK cells can persist and expand in vivo following adoptive transfer and may have a role in the treatment of late stage malignancies. NK also express an activating Fc receptor that mediates antibody-dependent cellular cytotoxicity (ADCC) and production of immune modulatory cytokines in response to antibody-coated targets. Nimotuzumab, an monoclonal antibody against EGFR (epidermal growth factor receptor), may enhance the ADCC effect of NK cell. This study will evaluate the safety of combination of nimotuzumab and NK Cell in treating advanced cancer patients. Blood samples will also be collected for research purposes.

DETAILED DESCRIPTION:
This is a phase I clinical study of expanded NK cells from autologous origin. The NK cell will be selected and expanded ex vivo and infused back into patients. Nimotuzumab will be used 24 hours before infusion. 21 advanced cancer patients are planned to receive two cycles of NK cells and Nimotuzumab treatment. Biomarkers and immunological markers are collected and analyzed as well.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed recurrent or metastatic cancer
2. Measurable disease
3. Progressed after all standard treatment
4. ECOG performance status of 0 to 2
5. Expected life span ≥ 3 months
6. Toxicities from prior treatment has resolved. Washout period is 4 weeks for chemotherapy, and 2 weeks for targeted therapy
7. Major organs function normally
8. Women at pregnant ages should be under contraception
9. Willing and able to provide informed consent

Exclusion Criteria:

1. Other malignancy within 5 years prior to entry into the study, expect for treated non melanoma skin cancer and cervical carcinoma in situ
2. Poor vasculature
3. Disease to the central nervous system
4. Blood-borne infectious disease, eg. hepatitis B
5. History of mandatory custody because of psychosis or other psychological disease inappropriate for treatment deemed by treating physician
6. With other immune diseases, or chronic use of immunosuppressants or steroids
7. Pregnancy (women of childbearing potential: Refusal or inability to use effective means of contraception)
8. Breastfeeding
9. Decision of unsuitableness by principal investigator or physician-in-charge

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-03-30 (Estimated); Study Completion 2019-11-27 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 6 month
  Number of Patients with Clinical or Biological Treatment-related Adverse Events and/or Dose Limiting Toxicities as a Measure of Safety and Tolerability of a Combination of Nimotuzumab and NK Cell as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Response Rate | 3 months
  Response will be evaluated according to RECIST v1.1

OTHER OUTCOMES:
Progression free survival (PFS) | 1 year
  From date of randomization until the date of first documented progression or date of death from any cause
Overall Survival (OS) | 1 year
  The time from randomization to death from any cause
Peripheral blood circulating tumor DNA | 6 weeks
  Peripheral circuiting tumor DNA is collected at baseline and 6 weeks after last treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shixiu Wu, Doctor, Principal Investigator — Hangzhou Cancer Hospital
Locations (1):
- Hangzhou Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No